CLINICAL TRIAL: NCT02936388
Title: A Randomized Phase II Trial of Transarterial Radioembolisation With Yttrium-90 (SIRT) in Comparison to Transarterial Chemoembolisation With Cisplatin (TACE) in Patients With Liver Metastases From Uveal Melanoma
Brief Title: Transarterial Radioembolisation in Comparison to Transarterial Chemoembolisation in Uveal Melanoma Liver Metastasis
Acronym: SirTac
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Caroline Anna Peuker, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SirTac2014
Record Dates: First submitted 2016-09-09; First posted 2016-10-18 (Estimated); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Uveal Melanoma
Keywords: uveal melanoma; liver metastasis; chemoembolisation; radioembolisation
MeSH Terms: conditions — Uveal Melanoma | interventions — Sirtuins; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): SIRT: Transarterial radioembolisation with Yttrium-90-bearing resin microspheres (SIR-Spheres®)
  Interventions: Procedure: SIRT
- Arm B (Active Comparator): DSM-TACE: Transarterial chemoembolisation with Cisplatin and EmboCept® S starch microspheres (PharmaCept GmbH)
  Interventions: Procedure: DSM-TACE

INTERVENTIONS:
Procedure: SIRT — catheter-based application of radioactive microspheres into the hepatic artery
  Other Names: Drug: Yttrium-90 microspheres (SIR-Spheres®)
  Arms: Arm A
Procedure: DSM-TACE — catheter-based application of chemotherapy and degradable starch microspheres into the hepatic artery
  Other Names: Drug: Cisplatin and EmboCept®
  Arms: Arm B

SUMMARY:
Characterisation of effect of SIRT and DSM-TACE as local treatment options for liver metastases in patients with advanced uveal melanoma with respect to progression-free survival and exploratory comparison of secondary endpoints regarding application, activity, adverse effects and impact on quality of life in a randomized study design.

DETAILED DESCRIPTION:
This is a randomized phase II trial to evaluate the effect of transarterial radioembolisation with yttrium-90 microspheres (SIRT) and transarterial chemoembolisation with cisplatin (DSM-TACE) in patients with liver metastases due to advanced uveal melanoma in terms of progression-free survival and multiple secondary endpoints.

Patients in study arm A will receive transarterial radioembolisation one time only. Patients in study arm B will receive transarterial chemoembolisation every 4 to 6 weeks until complete tumor devascularisation is observed or disease progression or intolerable toxicity occur. At the time of local tumor progression patients will be offered the other treatment respectively (either SIRT or DSM-TACE) as part of the study.

ELIGIBILITY:
Inclusion Criteria (main):

* ECOG Performance Status of 0, 1 or 2
* Histologically or cytologically confirmed liver metastases of uveal melanoma
* At least one measurable lesion according to RECIST criteria v1.1 determined MRI (if contraindications against MRI exist CT with contrast media can is allowed)
* Metastases in other sides are allowed if not in need of treatment (e.g. asymptomatic bone metastasis without indication for radiation)
* Prior treatment with systemic anti-cancer therapy is allowed if terminated ≥ 4 weeks prior to study treatment start and recovery from toxicity is achieved
* Surgery in general and hepatic surgery in particular (e.g. lobe resection, radiofrequency ablation) prior to study enrollment are allowed if realized ≥ 4 weeks prior to study enrollment and recovery from surgery is achieved

Exclusion Criteria (main):

* Surgically treatable liver metastases
* Previous intraarterial hepatic treatment (e.g. radioembolisation, chemoembolisation, intraarterial chemotherapy, isolated or percutaneous hepatic perfusion)
* Previous treatment with external liver radiation
* Major intrahepatic occlusion of the portal vein and/or tumor infiltration of the portal vein
* Liver cirrhosis Child-Pugh C
* Progressive liver failure
* Renale failure, bone marrow insufficiency, coagulopathy
* Uncontrolled or severe medical conditions which could impair the ability to participate in the trial such as unstable cardiac disease or uncontrolled infection
* Other malignancy and/or metastases in need of treatment
* Current treatment with any anti-cancer therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-01; Primary Completion 2024-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Pregression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Keilholz, Prof. Dr. med., Principal Investigator — Charité Universitätsmedizin Berlin, Charité Comprehensive Cancer Center (CCCC)
Locations (1):
- Charité - University Medicine Berlin, Dept. of Haematology, Medical Oncology and Tumor Immunology, Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Related Info — https://cccc.charite.de/forschung/klinische_studien/solide_tumorerkrankungen/leber_und_gallentumore_icd10_c22_c24/